CLINICAL TRIAL: NCT01896635
Title: Faecal Microbiota Transplantation for Chronic Active Ulcerative Colitis - A Randomised Double Blind Controlled Study of Efficacy & Safety
Brief Title: Faecal Microbiota Transplantation in Ulcerative Colitis
Acronym: FOCUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Dr. Sudarshan Paramsothy, Gastroenterologist / PhD candidate, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOCUS
Record Dates: First submitted 2013-07-06; First posted 2013-07-11 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease; Fecal Transplantation; Fecal Microbiota Transplantation
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- FMT infusions (Active Comparator): FMT infusions constituted from stool provided by healthy, screened donors
  Interventions: Biological: FMT infusions
- Placebo arm (Placebo Comparator): Placebo infusions
  Interventions: Other: Placebo infusion

INTERVENTIONS:
Biological: FMT infusions — Active FMT derived from healthy anonymous pre-screened donors
  Arms: FMT infusions
Other: Placebo infusion — Placebo infusion not containing any donor microbial material
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to determine whether fecal microbiota transplantation (FMT) is safe and efficacious in the treatment of chronic active ulcerative colitis (UC) by conducting a randomised controlled trial

DETAILED DESCRIPTION:
This study involves the assessment of the safety and efficacy of FMT in the treatment and induction of remission for patients with mild to moderate ulcerative colitis. It is a double blind study with patients randomised in a 1:1 manner to either active or placebo therapy

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis >3 months duration
* Active mild-moderate ulcerative colitis (Mayo 4-10)
* Ulcerative colitis of any extent except isolated proctitis < 5cm
* Live within driving distance of clinical site (to attend multiple study visits)

Exclusion Criteria:

* Pregnancy
* Active gastrointestinal infection
* Other gastrointestinal disease / comorbidities
* Prior colonic surgery
* Recent antibiotic or probiotic use
* Prednisone > 20mg
* Monoclonal antibody immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Composite Clinical remission & Endoscopic remission / response as measured by Mayo subscores | 8 weeks

SECONDARY OUTCOMES:
Clinical remission as measured by Mayo subscores | 8 weeks
Clinical response as measured by Mayo subscores | 8 weeks
Endoscopic healing as measured by UCEIS | 8 weeks
Treatment failure rate as defined by Mayo subscores | 8 weeks
Quality of life as measured by IBDQ | 8 weeks
Safety and tolerability as measured by adverse event data | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Mitchell, BSc PhD, Principal Investigator — University of New South Wales; Alissa Walsh, MBBS, Principal Investigator — St Vincent's Hospital, Sydney; Johan van den Bogaerde, MBChB PhD, Principal Investigator — Nambour General Hospital, Queensland; Douglas Samuel, MBBS MMed, Principal Investigator — Bankstown-Lidcombe Hospital, Sydney; Nadeem O Kaakoush, BSc PhD, Principal Investigator — University of New South Wales; Michael Kamm, MBBS MD, Principal Investigator — University of Melbourne
Locations (3):
- Australia (3):
  - St Vincent's Hospital, Sydney, New South Wales
  - Bankstown-Lidcombe Hospital, Sydney, New South Wales
  - Nambour General Hospital, Nambour, Queensland

REFERENCES:
- [Derived] Paramsothy S, Nielsen S, Kamm MA, Deshpande NP, Faith JJ, Clemente JC, Paramsothy R, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Lin E, Borody TJ, Wilkins MR, Colombel JF, Mitchell HM, Kaakoush NO. Specific Bacteria and Metabolites Associated With Response to Fecal Microbiota Transplantation in Patients With Ulcerative Colitis. Gastroenterology. 2019 Apr;156(5):1440-1454.e2. doi: 10.1053/j.gastro.2018.12.001. Epub 2018 Dec 6. PMID 30529583
- [Derived] Paramsothy S, Kamm MA, Kaakoush NO, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Paramsothy R, Xuan W, Lin E, Mitchell HM, Borody TJ. Multidonor intensive faecal microbiota transplantation for active ulcerative colitis: a randomised placebo-controlled trial. Lancet. 2017 Mar 25;389(10075):1218-1228. doi: 10.1016/S0140-6736(17)30182-4. Epub 2017 Feb 15. PMID 28214091
- [Derived] Paramsothy S, Walsh AJ, Borody T, Samuel D, van den Bogaerde J, Leong RW, Connor S, Ng W, Mitchell HM, Kaakoush NO, Kamm MA. Gastroenterologist perceptions of faecal microbiota transplantation. World J Gastroenterol. 2015 Oct 14;21(38):10907-14. doi: 10.3748/wjg.v21.i38.10907. PMID 26478682
- [Derived] Paramsothy S, Borody TJ, Lin E, Finlayson S, Walsh AJ, Samuel D, van den Bogaerde J, Leong RW, Connor S, Ng W, Mitchell HM, Kaakoush N, Kamm MA. Donor Recruitment for Fecal Microbiota Transplantation. Inflamm Bowel Dis. 2015 Jul;21(7):1600-6. doi: 10.1097/MIB.0000000000000405. PMID 26070003